CLINICAL TRIAL: NCT07351539
Title: Effects of Plyometric Training on Balance, Joint Position Sense, and Explosive Strength in Young Taekwondo Athletes
Brief Title: The Effects of Plyometric Training on Balance, Joint Position Sense, and Explosive Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ali Osman Kıvrak, Associate Professor, Selcuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SelcukU--SBF-AEB-AOK-2025-002
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Effects of Plyometric Training on Balance, Joint Position Sense, and Explosive Strength in Healthy Young Taekwondo Athletes
Keywords: Explosive Strength; Balance; Joint Position Sense; Plyometric Training; Taekwondo
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plyometric (Experimental): A total of 20 club-level taekwondo athletes aged between 15 and 18 years from Konya province voluntarily participated in the study. The participants were divided into two groups: an experimental group consisting of 10 athletes (5 female, 5 male) and a control group consisting of 10 athletes (5 female, 5 male). Inclusion criteria required that participants had no current injuries or any recent injuries that could adversely affect their performance. A pre-test-post-test research design was employed.
  Interventions: Other: Plyometric

INTERVENTIONS:
Other: Plyometric — A total of 20 club-level taekwondo athletes aged between 15 and 18 years from Konya province voluntarily participated in the study. The participants were divided into two groups: an experimental group consisting of 10 athletes (5 female, 5 male) and a control group consisting of 10 athletes (5 female, 5 male). Inclusion criteria required that participants had no current injuries or any recent injuries that could adversely affect their performance. A pre-test-post-test research design was employed. Following the measurement of anthropometric characteristics (height and body mass), assessments of balance, knee joint position sense, standing long jump, and vertical jump were conducted. After the completion of pre-test measurements, the experimental group performed a plyometric training program in addition to their regular taekwondo training for eight weeks, three times per week (Monday, Wednesday, and Friday), whereas the control group continued only their regular taekwondo training.

SUMMARY:
The purpose of this study was to investigate the effects of plyometric training on balance, joint position sense, and explosive strength in young taekwondo athletes.

A total of 20 taekwondo athletes aged between 15 and 18 years from Konya province voluntarily participated in the study. The participants were divided into two groups: an experimental group consisting of 10 athletes (5 female, 5 male) and a control group consisting of 10 athletes (5 female, 5 male). In addition to regular taekwondo training, the experimental group performed a plyometric training program three days per week for eight weeks, whereas the control group continued only their regular taekwondo training. Paired-sample and independent-sample t-tests were used for group comparisons.

DETAILED DESCRIPTION:
Methods:

Study design and participants A total of 20 club-level taekwondo athletes aged between 15 and 18 years from Konya province voluntarily participated in the study. The participants were divided into two groups: an experimental group consisting of 10 athletes (5 female, 5 male) and a control group consisting of 10 athletes (5 female, 5 male). Inclusion criteria required that participants had no current injuries or any recent injuries that could adversely affect their performance. A pre-test-post-test research design was employed. Following the measurement of anthropometric characteristics (height and body mass), assessments of balance, knee joint position sense, standing long jump, and vertical jump were conducted. After the completion of pre-test measurements, the experimental group performed a plyometric training program in addition to their regular taekwondo training for eight weeks, three times per week (Monday, Wednesday, and Friday), whereas the control group continued only their regular taekwondo training. Post-test measurements were obtained from both groups at the end of the eight-week training period. All assessments were conducted in the performance measurement laboratory of the Faculty of Sport Sciences.

Height Measurements The heights of the volunteer taekwondo athletes were recorded in centimeters (cm). To ensure accuracy and eliminate potential sources of error during height measurement, athletes were measured barefoot and wore only a t-shirt and shorts. Measurements were conducted using an MST-B01 stadiometer with a precision of 0.01 mm.

Body Weight Measurements Measurements were taken twice, as the first and second assessments, using the Tanita BC 601 body composition analyzer. Care was taken to ensure that the device was placed on a flat and hard surface during the measurements. Athletes were barefoot and wore no clothing that could affect their weight. Body weights were recorded in kilograms (kg).

Balance Test Balance performance was assessed using the Biodex Balance System (Biodex Balance System, BBS; Biodex Medical Systems Inc., Shirley, NY, USA). The system consists of a movable balance platform capable of tilting up to 20° in all directions, allowing a 360° range of motion. The device provides 12 adjustable stability levels, with Level 1 representing the least stable and Level 12 the most stable condition. The platform is connected to dedicated computer software that enables objective evaluation of balance performance, providing an overall postural stability index as well as directional indices in the anteroposterior (AP) and mediolateral (ML) planes. The postural stability index reflects overall balance ability, with higher scores indicating poorer balance performance. Prior to testing, participants were asked to identify their dominant leg. After determining leg dominance, athletes were positioned on the platform standing on the dominant leg with the knee slightly flexed at approximately 45°, while the non-dominant leg was flexed at 90° at the knee. Participants maintained their arms crossed over the chest throughout the test. During the assessment, visual feedback from the screen was eliminated, and athletes were instructed to focus on a fixed point located approximately 1 m away at eye level. For postural control assessment, the platform stability was set at Level 8 under eyes-open (EO) conditions and Level 10 under eyes-closed (EC) conditions. Measurements were conducted under both EO and EC conditions. Before formal testing, participants performed three familiarization trials, each lasting 30 s. Subsequently, balance tests were conducted eight times under EO and EC conditions (including normal balance, balance during a mental task, balance during a visual task, and balance during a verbal task), with each trial lasting 30 s. A 5-min rest interval was provided between tests. Pre- and post-training measurements were administered using identical testing procedures.

Knee Joint Position Sense Assessment Knee joint position sense was assessed using an isokinetic dynamometer (HUMAC NORM, Lumex Inc., Ronkonkoma, NY, USA). Prior to testing, the dynamometer settings were individually adjusted according to each participant's anthropometric characteristics. Measurements were performed for both the dominant and non-dominant legs. Participants were provided with three familiarization trials before data collection to ensure adaptation to the isokinetic dynamometer. During testing, the knee joint of both the dominant and non-dominant limbs was positioned at maximum flexion and then slowly moved toward extension. At flexion angles of 30°, 45°, and 60°, the movement was paused for 10 s at each angle to allow participants to learn the target positions. Subsequently, the knee was returned to maximum flexion, and participants were instructed to actively reproduce the previously learned target angles (30°, 45°, and 60°) by extending the knee. Each angle was tested three times for both the dominant and non-dominant legs. A 2-min rest period was provided between trials. The mean absolute error from the target angles was calculated, and the average deviation was recorded as the knee joint position sense value for both the dominant and non-dominant legs.

Vertical Jump Test Vertical jump performance was assessed using a TKK 5406 jump meter. Prior to testing, participants were allowed sufficient practice trials to become familiar with the testing device. During the test, athletes stood on the measurement mat with both feet and were instructed to jump as high as possible at a self-selected time following the visual signal from the device. Arm and leg swing were permitted during the jump. Participants were instructed to land on the mat with both feet simultaneously after the jump. Vertical jump height was displayed on the device screen and recorded immediately after each trial. The test was repeated three times with a 1-min rest interval between trials. The highest value obtained from the three trials was recorded as the participant's vertical jump performance.

Standing Long Jump Test Athletes were positioned with their toes just behind the starting line, feet at a normal width, and with their arms extended forward and knees bent in a pre-jump stance. They were instructed to jump as far as possible, using their arms for momentum, and both feet were to land simultaneously. The distance from the starting line to the athlete's heels was measured in centimeters and recorded. Athletes were given two attempts, and the best result was taken for analysis.

Statistical Analysis Data analysis was performed using the SPSS software (Version 27.0). Descriptive statistics were used to summarize all quantitative data and are presented as mean and standard deviation. The normality of data distribution was assessed using the Shapiro-Wilk test. Based on the assumption of normal distribution, independent-samples t-tests were applied to compare the two independent groups, while paired-samples t-tests were used to compare pre-test and post-test measurements within the same group. The level of statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

• When forming the groups, care was taken to ensure that none of the athletes were currently undergoing injury rehabilitation or had any recent injuries that could affect their performance. Additionally, all voluntary participants underwent health screening to verify their current health status.

Exclusion Criteria:

• Athletes with injuries or illnesses were not included in the study.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Balance Test | [Time Frame: For 8 weeks from the start of the study]
  After determining leg dominance, athletes were positioned on the platform standing on the dominant leg with the knee slightly flexed at approximately 45°, while the non-dominant leg was flexed at 90° at the knee. Participants maintained their arms crossed over the chest throughout the test. During the assessment, visual feedback from the screen was eliminated, and athletes were instructed to focus on a fixed point located approximately 1 m away at eye level. For postural control assessment, the platform stability was set at Level 8 under eyes-open (EO) conditions and Level 10 under eyes-closed (EC) conditions. Measurements were conducted under both EO and EC conditions. Before formal testing, participants performed three familiarization trials, each lasting 30 s. Subsequently, balance tests were conducted eight times under EO and EC conditions, with each trial lasting 30 s. A 5-min rest interval was provided between tests.
Knee Joint Position Sense Assessment | [Time Frame: For 8 weeks from the start of the study]
  Participants were provided with three familiarization trials before data collection to ensure adaptation to the isokinetic dynamometer. During testing, the knee joint of both the dominant and non-dominant limbs was positioned at maximum flexion and then slowly moved toward extension. At flexion angles of 30°, 45°, and 60°, the movement was paused for 10 s at each angle to allow participants to learn the target positions. Subsequently, the knee was returned to maximum flexion, and participants were instructed to actively reproduce the previously learned target angles (30°, 45°, and 60°) by extending the knee. Each angle was tested three times for both the dominant and non-dominant legs. A 2-min rest period was provided between trials. The mean absolute error from the target angles was calculated, and the average deviation was recorded as the knee joint position sense value for both the dominant and non-dominant legs.
Vertical Jump Test | [Time Frame: For 8 weeks from the start of the study]
  Vertical jump performance was assessed using a TKK 5406 jump meter. Prior to testing, participants were allowed sufficient practice trials to become familiar with the testing device. During the test, athletes stood on the measurement mat with both feet and were instructed to jump as high as possible at a self-selected time following the visual signal from the device. Arm and leg swing were permitted during the jump. Participants were instructed to land on the mat with both feet simultaneously after the jump. Vertical jump height was displayed on the device screen and recorded immediately after each trial. The test was repeated three times with a 1-min rest interval between trials. The highest value obtained from the three trials was recorded as the participant's vertical jump performance.
Standing Long Jump Test | [Time Frame: For 8 weeks from the start of the study]
  Athletes were positioned with their toes just behind the starting line, feet at a normal width, and with their arms extended forward and knees bent in a pre-jump stance. They were instructed to jump as far as possible, using their arms for momentum, and both feet were to land simultaneously. The distance from the starting line to the athlete's heels was measured in centimeters and recorded. Athletes were given two attempts, and the best result was taken for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Osman Kıvrak, Associate Professor, Principal Investigator — Department of Coaching Education, Faculty of Sport Sciences, Selçuk University; Ahmet Mücahit Özcan, MSc, Principal Investigator — Department of Coaching Education, Faculty of Sport Sciences, Selçuk University
Locations (1):
- Alaeddin Keykubat Yerleşkesi Akademi Mah. Yeni İstanbul Cad. Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided